CLINICAL TRIAL: NCT05569772
Title: Semaglutide for the Treatment of Glucose Intolerance in Women with Prior Gestational Diabetes: a Double Blind RCT
Brief Title: Semaglutide for the Treatment of Glucose Intolerance in Women with Prior Gestational Diabetes
Acronym: SERENA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); Universitair Ziekenhuis Brussel (Other); General Hospital Groeninge (Other); Onze Lieve Vrouw Hospital (Other); Jessa Hospital (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Vitaz (Other); Centre Hospitalier Universitaire de Liege (Other); Erasme University Hospital (Other); Centre Hospitalier Mouscron (Unknown); Jan Yperman Ziekenhuis (Other); AZ Turnhout (Other); AZ Sint-Lucas Brugge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S66967; 2022-502082-22-00 (Other: EU CT number)
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Glucose Intolerance After a Recent History of Gestational Diabetes
Keywords: gestational diabetes; glucose intolerance postpartum; prevention; type 2 diabetes; GLP-1 agonist; semaglutide
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: multi-centric double blind RCT
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide (Active Comparator): semaglutide SC once weekly, up titration over 2 month period to 1mg/week (0.25mg once weekly, after 4 weeks 0.5mg once weekly and after 8 weeks the maintenance dose of 1mg once weekly), treatment duration of max. 3 years
  Interventions: Drug: Semaglutide Pen Injector
- placebo (Placebo Comparator): placebo SC once weekly, the same dose-escalation regimen, using matching injections, treatment duration of max. 3 years
  Interventions: Drug: Semaglutide placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — maintenance dose of 1mg SC once weekly
  Other Names: Ozempic
  Arms: semaglutide
Drug: Semaglutide placebo — maintenance dose of 1mg SC once weekly
  Arms: placebo

SUMMARY:
Gestational diabetes (GDM) is an important contributor to the increasing prevalence of type 2 diabetes (T2DM). Women with glucose intolerance in early postpartum are a particularly high-risk group with about 50% who will develop T2DM within 5 years after the delivery. Moreover, women with a history of GDM progress more rapidly to T2DM compared to women with similarly elevated glucose levels. Early intervention after the index pregnancy is therefore crucial to prevent T2DM. With the SERENA project, the investigators aim to reduce the risk to develop T2DM with the long-acting GLP-1 agonist semaglutide in women with a recent history of GDM and glucose intolerance in early postpartum.

DETAILED DESCRIPTION:
Patient population: Women with a recent history of gestational diabetes (GDM) and persistent glucose intolerance in early postpartum are a particularly high risk group, with about 50% developing type 2 diabetes (T2DM) within 5 years after the delivery. Semaglutide is a long-acting glucagon-like peptide-1 (GLP-1) agonist with multiple beneficial metabolic effects, including glucose lowering effect, weight loss and cardiovascular protective effects. The investigators hypothesize that in women with prior GDM and glucose intolerance in early postpartum, treatment with semaglutide will reduce the risk to develop T2DM on the long-term compared to placebo.

Intervention and comparison: Belgian multi-centric double blind RCT with 13 centers to compare semaglutide (once weekly) with placebo in women with a recent history of GDM and glucose intolerance [impaired fasting glycaemia (IFG) and/or impaired glucose tolerance (IGT)] 6-24 weeks postpartum. Participants will be 1/1 randomized to semaglutide or placebo on a background of lifestyle measures. Semaglutide will be uptitrated to 1mg/week over a 8-week period. Participants will be followed-up for 3 years. Participants will receive a 75g oral glucose tolerance test (OGTT) 3-6 months after the stop of the intervention. Randomization will be stratified according to BMI at the early postpartum visit (<25; 25-29.9 and ≥30Kg/m²).

Outcomes: The primary endpoint is the development of T2DM by 160 weeks defined by fasting glycaemia, OGTT and/or HbA1c according to the ADA criteria. Important secondary endpoints include the need for rescue therapy for diabetes, regression to normoglycaemia, weight loss, beta-cell function, insulin resistance and the metabolic syndrome. To achieve 80% power, we plan a sample size of 252 to detect an estimated 50% reduction in the risk to develop T2DM between both groups, assuming a 30% loss to follow-up during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control
3. History of GDM (diagnosed with 2013 WHO criteria 24-32 weeks of pregnancy) and glucose intolerance 6-24 weeks postpartum (based on the ADA criteria)
4. Needs to be able to understand and speak Dutch, French or English

Exclusion Criteria:

* 1. Participant has a history of any type of diabetes or auto-antibodies for type 1 diabetes, history of pancreatitis, family or personal history of medullary thyroid carcinoma or personal history of thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, severe psychiatric disorder in the past year, heart failure NYHA class 4, end-stage renal disease (eGFR <15) or dialysis, or history of bariatric surgery 2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol 3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial 4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive 5. Participation in an interventional Trial with an investigational medicinal product or device 6. Age <18 years, breastfeeding >24 weeks postpartum or HbA1c≥6.5% at the time of the OGTT in pregnancy 7. Use of medication with significant impact on glycaemia (such as high dose glucocorticoids or metformin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
type 2 diabetes | by 160 weeks
  development of type 2 diabetes defined by fasting glycaemia, oral glucose tolerance test and/or HbA1c according to the ADA criteria

SECONDARY OUTCOMES:
medication for diabetes | by 160 weeks
  percentage need for rescue therapy for diabetes
prediabetes | by 160 weeks
  percentage prediabetes based on fasting glycaemia, oral glucose tolerance test and/or HbA1c (ADA criteria)
normoglycaemia | by 160 weeks
  percentage regression to normoglycaemia, based on fasting glycaemia, oral glucose tolerance test and/or HbA1c (ADA criteria)
BMI | by 160 weeks
  mean BMI (Kg/m2)
waist circumference | by 160 weeks
  mean waist circumference (cm)
waist/hip ratio | by 160 weeks
  waist/hip circumference ratio
5% weight loss | by 160 weeks
  percentage weight loss ≥5%
10% weight loss | by 160 weeks
  percentage weight loss ≥10%
15% weight loss | by 160 weeks
  percentage weight loss ≥15%
body fat percentage | by 160 weeks
  percentage body fat measured by bioelectrical impedance analysis
HOMA-B index | by 160 weeks
  Beta-cell function measured by the HOMA-B index
insulinogenic index | by 160 weeks
  Beta-cell function measured by the by the insulinogenic index divided by HOMA-insulin resistance index
ISSI-2 index | by 160 weeks
  Beta-cell function measured by theby the insulin-secretion sensitivity-2 index
the Stumvoll index. | by 160 weeks
  Beta-cell function measured by the Stumvoll index.
Matsuda index | by 160 weeks
  whole body Insulin sensitivity measured by the insulin sensitivity index of Matsuda
HOMA-IR | by 160 weeks
  the reciprocal of the homeostasis model assessment of insulin resistance (1/HOMA-IR)
metabolic syndrome | by 160 weeks
  percentage of the metabolic syndrome based on the WHO criteria
Hypertension | by 160 weeks
  percentage blood pressure ≥140/90mmHg
heart rate | by 160 weeks
  mean heart rate
LDL cholesterol | by 160 weeks
  percentage LDL cholesterol ≥100mg/dl
Triglycerides | by 160 weeks
  percentage triglycerides ≥150mg/dl
hypoglycaemia | by 160 weeks
  percentage with hypoglycaemia (<54mg/dl)
gastro-intestinal side effects | by 160 weeks
  percentage nausea, vomiting or diarrhea
self-reported quality of life | by 160 weeks
  health-related quality of life by SF-36 questionnaire
symptoms of depression | by 160 weeks
  the 20-item Center for Epidemiologic Studies-Depression (CES-D) questionnaire
anxiety | by 160 weeks
  six-item short-form of the State-Trait Anxiety Inventory questionnaire on anxiety (STAI)
Diabetes risk perception | by 160 weeks
  Diabetes Risk perception questionnaire, a validated questionnaire to evaluate the perception to develop diabetes
sleep quality | by 160 weeks
  The validated Pittsburg sleep quality index to evaluate sleep quality
diabetes remission | by 172-184 weeks (3-6 months after end of therapy)
  diabetes remission rate after treatment stop, defined by fasting, OGTT and/or HbA1c

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (13):
  - OLV-Aalst-Asse, Aalst
  - UZA, Antwerp
  - ZNA,, Antwerp
  - AZ St Jan Brugge, Bruges
  - Erasme, Brussels
  - UZ Brussel, Brussels
  - Jan Yperman, Ieper
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - Centre Hospitalier Mouscron, Mouscron
  - Vitaz, Sint-Niklaas
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No